CLINICAL TRIAL: NCT07078539
Title: Comparative Effect of Kaltenborn and Mulligan Mobilization With Intrinsic Foot Muscle Strengthening on Pain, Functional Status, and Windlass Mechanism in Patients With Plantar Fasciitis
Brief Title: Effect of Kaltenborn vs Mulligan Mobilization With Intrinsic Foot Strengthening in Plantar Fasciitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0164 -Adeena
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Plantar Fascitis; Heel Pain Syndrome
Keywords: Manual Therapy; Intrinsic Foot Muscle Strengthening; Heel Pain; Kaltenborn Mobilization; Mulligan Mobilization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kaltenborn Mobilization Group (Experimental): Participants in this group will receive Kaltenborn mobilization techniques applied to the talocrural and subtalar joints. Mobilizations will be performed as Grade III passive accessory glides for 10 repetitions per joint, each sustained for 15 seconds with a 10-second rest interval
  Interventions: Other: Kaltenborn Mobilization Group
- Mulligan Mobilization Group (Experimental): Participants in this group will receive Mulligan mobilization with movement (MWM) techniques applied to the talocrural and subtalar joints. Mobilizations will be applied as 3 sets of 10 repetitions per joint with 1-minute rest between sets.
  Interventions: Other: Mulligan Mobilization Group

INTERVENTIONS:
Other: Kaltenborn Mobilization Group — Participants in this group will receive Kaltenborn mobilization techniques applied to the talocrural and subtalar joints. Mobilizations will be performed as Grade III passive accessory glides for 10 repetitions per joint, each sustained for 15 seconds with a 10-second rest interval
  Conventional treatment includs therapeutic ultrasound (3 MHz, 1.5 W/cm², continuous mode for 5 minutes), plantar fascia and calf stretching (10 minutes, 1 set of 10 reps), intrinsic foot muscle strengthening exercises (toe curls and towel curls for 10 minutes, 2 sets of 10 reps), and cryotherapy at home for 10 minutes daily. The intervention will be delivered twice weekly for 3 weeks.
  Arms: Kaltenborn Mobilization Group
Other: Mulligan Mobilization Group — Participants in this group will receive Mulligan mobilization with movement (MWM) techniques applied to the talocrural and subtalar joints. Mobilizations will be applied as 3 sets of 10 repetitions per joint with 1-minute rest between sets.
  Conventional treatment includs therapeutic ultrasound (3 MHz, 1.5 W/cm², continuous mode for 5 minutes), plantar fascia and calf stretching (10 minutes, 1 set of 10 reps), intrinsic foot muscle strengthening exercises (toe curls and towel curls for 10 minutes, 2 sets of 10 reps), and cryotherapy at home for 10 minutes daily. The intervention will be delivered twice weekly for 3 weeks.
  Arms: Mulligan Mobilization Group

SUMMARY:
This study will compare the effects of Kaltenborn and Mulligan ankle mobilization techniques, combined with intrinsic foot muscle strengthening, on pain, functional status, and dorsiflexion range of motion in patients with plantar fasciitis. Eighty-two participants with chronic heel pain will be randomly allocated into two groups. Both groups will receive standard care including ultrasound therapy, stretching, and cryotherapy, while Group A will receive Kaltenborn mobilization and Group B will receive Mulligan mobilization. Pain, function, and ankle range of motion will be assessed at baseline and after three weeks of treatment.

DETAILED DESCRIPTION:
This prospective randomized clinical trial will aim to evaluate and compare the effectiveness of two manual therapy techniques-Kaltenborn and Mulligan mobilizations-combined with intrinsic foot muscle strengthening in the treatment of plantar fasciitis. The study will be conducted at two physiotherapy clinics in Sialkot, Pakistan. A total of 82 eligible participants aged 30-60 years, diagnosed with plantar fasciitis, will be enrolled using non-probability convenience sampling and then randomised into two equal groups through the lottery method.

Group A will receive Kaltenborn mobilization techniques applied to the talocrural and subtalar joints, in addition to conventional treatment (therapeutic ultrasound, plantar fascia and calf stretching, intrinsic foot muscle strengthening, and cryotherapy). Group B will receive Mulligan mobilization with movement (MWM) applied to the same joints, alongside the same conventional treatment.

Interventions will be delivered twice weekly for three weeks (total six sessions). The primary outcomes will include changes in pain intensity (Numeric Pain Rating Scale), functional disability (Foot Function Index), and ankle dorsiflexion range of motion (measured using a goniometer). Measurements will be taken at baseline and at the end of the third week. It is hypothesised that Kaltenborn mobilization may demonstrate superior outcomes in pain reduction and functional improvement compared to Mulligan MWM when combined with strengthening exercises.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 30-60.

  * Both genders (male and female) included.
  * Subjects with the ankle and heel pain complain especially morning or after rest and limited ankle ROM due to pain
  * Positive Windlass test: Pain increase upon toe standing and decreases upon walking.

Duration of pain in 4 weeks or more.

* Tenderness on medial calcaneal tuberosity.
* NPRS score of 4 or more

Exclusion Criteria:

* Patients contraindicated to manual therapy (tumor, fracture or osteoporosis). Any history of knee, tibia, fibula, ankle or foot surgery or stress fracture of calcaneum.

  * Previously received physiotherapy treat.
  * History of non-steroidal anti-inflammatory medications or corticosteroid injection in last 3 weeks prior to surgery.
  * Pregnancy (because of sudden weight changes and pedal edema which causes heel pain).
  * Conditions like rheumatoid arthritis, ankylosing spondylitis, systematic lupus erythematous, peripheral neuropathy, sever's disease, severe vascular disease or tarsal tunnel.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Baseline and at the end of Week 3 (post-intervention)
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), a validated 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain).
Foot Function Index - FFI | Baseline and at the end of Week 3 (post-intervention)
  Functional disability will be evaluated using the Foot Function Index (FFI), a validated questionnaire assessing foot pain, disability, and activity limitation. It comprises 23 items scored on a visual analogue scale, with higher scores indicating greater impairment.
Ankle Dorsiflexion Range of Motion | Baseline and at the end of Week 3 (post-intervention)
  Ankle dorsiflexion will be measured using a universal goniometer to assess changes in passive range of motion.
Windlass Test | Baseline and at the end of Week 3 (post-intervention)
  The Windlass Test will be used as a clinical indicator of plantar fascia integrity and responsiveness. The test will be performed in a weight-bearing position by passively dorsiflexing the great toe while the patient stands on the affected foot. A positive result is defined by reproduction of heel or arch pain during the manoeuvre.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Zia, Phd Scholar, Principal Investigator — Riphah International University / Mayo Hospital, Lahore; Adeena Nazim, MSc Student, Principal Investigator — Riphah International University
Locations (1):
- Bashir Health Services, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szajkowski S, Pasek J, Cieslar G. Dose Escalation Can Enhance the Therapeutic Potential of Radial Extracorporeal Shock-Wave Therapy in the Treatment of Plantar Fasciitis in Runners. Medicina (Kaunas). 2024 May 6;60(5):766. doi: 10.3390/medicina60050766. PMID 38792948
- [Background] Boob MA Jr, Phansopkar P, Somaiya KJ. Physiotherapeutic Interventions for Individuals Suffering From Plantar Fasciitis: A Systematic Review. Cureus. 2023 Jul 31;15(7):e42740. doi: 10.7759/cureus.42740. eCollection 2023 Jul. PMID 37654968
- [Background] Rathleff MS, Molgaard CM, Fredberg U, Kaalund S, Andersen KB, Jensen TT, Aaskov S, Olesen JL. High-load strength training improves outcome in patients with plantar fasciitis: A randomized controlled trial with 12-month follow-up. Scand J Med Sci Sports. 2015 Jun;25(3):e292-300. doi: 10.1111/sms.12313. Epub 2014 Aug 21. PMID 25145882
- [Background] Maheta U, Thakarar S, Thakarar J, Pandita V, Patel SB, Ranu A, et al. EFFECTIVENESS OF MAITLAND MOBILIZATION VERSUS MULLIGAN MOBILIZATION FOR FLATFOOT IN THE MIDTARSAL JOINT.
- [Background] Shabbir S, Ahmad A, Munawar A, Siddique K, Perwaiz S. Comparison of mobilization with movement and dorsiflexion night splint with and without routine exercises in patients with plantar fasciitis. Rawal Medical Journal. 2022;47(3):650-.